CLINICAL TRIAL: NCT02708498
Title: Implementation of Knowledge-Based Palliative Care for Frail Older Persons in Nursing Homes
Brief Title: Implementation of Knowledge-Based Palliative Care
Acronym: KUPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Linnaeus University (Other); The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-2759; 2014-0071 (Other Grant/Funding Number: The Vardal Foundation)
Record Dates: First submitted 2016-02-26; First posted 2016-03-15 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Ageing
Keywords: Palliative care; Frail elderly; Comorbidity; Staff Development; Nursing Homes
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: The knowledge-based palliative care intervention was conducted as a non-randomized control trial.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Kronoberg Educational Intervention (Experimental): The educational intervention is provided to ten nursing homes.
  Interventions: Behavioral: Educational Intervention
- Skåne Control (No Intervention): The control group consists of an equal number of nursing homes. This group receives no intervention.
- Skåne Educational Intervention (Experimental): The educational intervention is provided to ten nursing homes.
  Interventions: Behavioral: Educational Intervention
- Kronoberg Control (No Intervention): The control group consists of an equal number of nursing homes. This group receives no intervention.

INTERVENTIONS:
Behavioral: Educational Intervention — The seminar groups will be led by two experienced clinical nurses and researchers from the field of palliative care and geriatric care. The educational material consist of six themes; values in palliative care, symptom relief, dignity and a dignified death, collaborative co-creating care, support to next of kin and dialogue with older persons and next of kin about death and dying. The content of the different themes will have a common core for each nursing home but will be adjusted based on the expressed needs of each nursing home. New themes can be created related to the needs of the unique nursing home. The participants in the seminar groups will reflect together over the content of the developed binder of educational material and will relate it to their own work in order to identify areas suitable for changes and/or development.
  Arms: Kronoberg Educational Intervention; Skåne Educational Intervention

SUMMARY:
The research on ageing during the last couple of decades has increasingly focused on questions regarding the quality of life and life satisfaction of the old people. Yet the research indicates that when it comes to the final stage of life, the end includes unnecessary suffering and the quality of life drops. Palliative care has traditionally been provided successfully to younger persons dying from incurable illnesses while older people dying of multiple morbidities or "old age" has received far less of this type of care. However, sixty percent of all people who died in Sweden in 2010 were at least 80 years old and it is well known that dying among older people often is a prolonged period of suffering. One reason might be that it is more difficult to identify when the final stages of life begins for older persons.

The purpose of this project is to implement and evaluate how a knowledge-based model for palliative care in nursing homes affects the quality of life and the participation in the care process for older persons in nursing homes and their next of kin. A second aim is to explore the staff's implementation process of palliative care and the role of the leadership. The final aim is to investigate which factors (barriers and facilitators) that affect the implementation process of this model.

DETAILED DESCRIPTION:
The project was planned to be conducted using a cross-over design in two counties in south of Sweden based on a feasibility/pilot study that was conducted during fall 2014 co-created palliative care educational intervention through seminars for professionals in nursing homes. Due to a more significant amount of drop-outs compared with expected (and for not receiving the total amount of applied foundation), the plan needed to be revised. The knowledge-based palliative care intervention was conducted as a non-blinded control trial, implemented over a six-month period in 30 nursing homes in two different counties in the south of Sweden (County A and County B). The data collection was made in two sequential periods in each county. First, the intervention was implemented in ten nursing homes in County A (Kronoberg County from April 2015), while ten nursing homes in County B served as a control group. Then, County B implemented the intervention (Skåne county from April 2016), and ten new nursing homes in County A, which had not received the intervention, were chosen as a control group. After the two sequential time periods were data from one intervention and one control group analysed. The selection through voluntary participation resulted in a mixture of both larger and smaller nursing homes in the two counties, as well as both from urban and rural areas.

Every seminar group met once a month and included different professions (unit manager, district nurse, assistant nurse, and other staff i.e. occupational therapist and physiotherapist). There were 5 meetings in each nursing home during a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Older persons living in the participating nursing homes
* Next of kin to older persons living in the participating nursing homes
* Staff working at the participating nursing homes
* Managers working at the participating nursing homes
* The participating nursing homes must be located in either Kronoberg County or Skåne County in Sweden

Exclusion Criteria:

* Not being cognitive able to participate in interviews or answering the questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1151 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Ahlström, PhD, Principal Investigator — Department of Health Sciences, Lund University
Locations (30):
- Sweden (30):
  - Bryggaren, Alvesta, Kronoberg County
  - Högåsen, Alvesta, Kronoberg County
  - Älmegården, Älmeboda, Kronoberg County
  - Asken, Grimslöv, Kronoberg County
  - Kvarngården, Ingelstad, Kronoberg County
  - Konga Allhus, Konga, Kronoberg County
  - Åbrinken, Lagan, Kronoberg County
  - Ljungberga, Ljungby, Kronoberg County
  - Ljungsätra, Ljungby, Kronoberg County
  - Brunnsgården, Ljungby, Kronoberg County
  - Torsgården, Lönashult, Kronoberg County
  - Furuliden, Moheda, Kronoberg County
  - Solängen, Ryd, Kronoberg County
  - Örnen, Tingsryd, Kronoberg County
  - Äppelgården, Urshult, Kronoberg County
  - Birkagården, Vaxjo, Kronoberg County
  - Hovslund, Vaxjo, Kronoberg County
  - Evelid, Vaxjo, Kronoberg County
  - Solhaga, Väckelsång, Kronoberg County
  - Björkliden, Vislanda, Kronoberg County
  - Skogsgläntan, Höör, Skåne County
  - Åsgården, Kågeröd, Skåne County
  - Mårtenslund, Lund, Skåne County
  - Brunnslyckan, Lund, Skåne County
  - Norrdala, Lund, Skåne County
  - Rönnebacken, Osby, Skåne County
  - Fästan, Södra Sandby, Skåne County
  - Solgården, Svalöv, Skåne County
  - Holmagården, Svedala, Skåne County
  - Ängslyckan, Teckomatorp, Skåne County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Persson HA, Ahlstrom G, Ekwall A. Professionals readiness for change to knowledge-based palliative care at nursing homes: a qualitative follow-up study after an educational intervention. BMC Palliat Care. 2022 Jul 20;21(1):132. doi: 10.1186/s12904-022-01018-y. PMID 35854375
- [Derived] Ahlstrom G, Rosen H, Persson EI. Quality of Life among Next of Kin of Frail Older People in Nursing Homes: An Interview Study after an Educational Intervention concerning Palliative Care. Int J Environ Res Public Health. 2022 Feb 24;19(5):2648. doi: 10.3390/ijerph19052648. PMID 35270339
- [Derived] Bokberg C, Sandberg J. Until death do us part Adult children's perspective of their parents' transition from living at home to moving into a nursing home and the time after death. BMC Geriatr. 2021 Nov 27;21(1):666. doi: 10.1186/s12877-021-02633-9. PMID 34837994
- [Derived] Sandgren A, Arnoldsson L, Lagerholm A, Bokberg C. Quality of life among frail older persons (65+ years) in nursing homes: A cross-sectional study. Nurs Open. 2021 May;8(3):1232-1242. doi: 10.1002/nop2.739. Epub 2020 Dec 13. PMID 34482652
- [Derived] Westergren A, Ahlstrom G, Persson M, Behm L. Next of kin participation in the care of older persons in nursing homes: A pre-post non-randomised educational evaluation, using within-group and individual person-level comparisons. PLoS One. 2021 Jan 25;16(1):e0244600. doi: 10.1371/journal.pone.0244600. eCollection 2021. PMID 33493153
- [Derived] Tjernberg J, Bokberg C. Older persons' thoughts about death and dying and their experiences of care in end-of-life: a qualitative study. BMC Nurs. 2020 Dec 16;19(1):123. doi: 10.1186/s12912-020-00514-x. PMID 33327960
- [Derived] Rosen H, Ahlstrom G, Lexen A. Psychometric properties of the WHOQOL-BREF among next of kin to older persons in nursing homes. Health Qual Life Outcomes. 2020 Apr 19;18(1):103. doi: 10.1186/s12955-020-01345-9. PMID 32306965
- [Derived] Westergren A, Behm L, Lindhardt T, Persson M, Ahlstrom G. Measuring next of kin's experience of participation in the care of older people in nursing homes. PLoS One. 2020 Jan 31;15(1):e0228379. doi: 10.1371/journal.pone.0228379. eCollection 2020. PMID 32004352
- [Derived] Rosen H, Behm L, Wallerstedt B, Ahlstrom G. Being the next of kin of an older person living in a nursing home: an interview study about quality of life. BMC Geriatr. 2019 Nov 21;19(1):324. doi: 10.1186/s12877-019-1343-4. PMID 31752709
- [Derived] Bokberg C, Behm L, Ahlstrom G. Next of kin's quality of life before and after implementation of a knowledge-based palliative care intervention in nursing homes. Qual Life Res. 2019 Dec;28(12):3293-3301. doi: 10.1007/s11136-019-02268-9. Epub 2019 Aug 14. PMID 31414348
- [Derived] Bokberg C, Behm L, Wallerstedt B, Ahlstrom G. Evaluation of person-centeredness in nursing homes after a palliative care intervention: pre- and post-test experimental design. BMC Palliat Care. 2019 May 31;18(1):44. doi: 10.1186/s12904-019-0431-8. PMID 31151438
- [Derived] Ahlstrom G, Nilsen P, Benzein E, Behm L, Wallerstedt B, Persson M, Sandgren A. Implementation of knowledge-based palliative care in nursing homes and pre-post post evaluation by cross-over design: a study protocol. BMC Palliat Care. 2018 Mar 22;17(1):52. doi: 10.1186/s12904-018-0308-2. PMID 29566688
- See also: The Swedish national knowledge support document for good palliative care — https://www.socialstyrelsen.se/globalassets/sharepoint-dokument/artikelkatalog/kunskapsstod/2013-6-4.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group Older People; Control Group Older People: Older persons: The inclusion criteria for the older persons were ≥ 65 years without dementia and with enough energy to manage a structured interview during up to one hour.
- Intervention Group Next-of-Kin; Control Group Next-of-kin: The next of kin: The inclusion criterion was someone who had a relation to one of the older persons living at the participating nursing homes but not necessarily family members or relatives.
- Intervention Group Staff; Control Group Staff: Staff: The inclusion criterion was staff at nursing homes (commonly assistant nurses, nurses, occupational therapists and physiotherapists).
- Intervention Group Managers: Managers: Managers at different levels with responsibility for the care and social service at the included nursing homes.
- Intervention Focus Groups: The focus groups took place at the intervention nursing homes and included 48 staff divided into six groups.
Period: Overall Study
Arm/Group | Intervention Group Older People | Control Group Older People | Intervention Group Next-of-Kin | Control Group Next-of-kin | Intervention Group Staff | Control Group Staff | Intervention Group Managers | Intervention Focus Groups
Started | 42 | 40 | 152 | 156 | 363 | 330 | 20 | 48
Completed | 22 | 21 | 90 | 105 | 167 | 198 | 20 | 48
Not Completed | 20 | 19 | 62 | 51 | 196 | 132 | 0 | 0
Not completed — Death | 20 | 19 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Unknown reason, missing data | 0 | 0 | 62 | 51 | 195 | 132 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Focus Groups Staff: The focus groups took place at the intervention nursing homes and included 40 staff divided into six groups.
- Total: Total of all reporting groups
Arm/Group | Intervention Group Older People | Control Group Older People | Intervention Group Next-of-Kin | Control Group Next-of-kin | Intervention Group Staff | Control Group Staff | Intervention Group Managers | Intervention Focus Groups Staff | Total
Number analyzed (Participants) | 42 | 40 | 152 | 156 | 363 | 330 | 20 | 48 | 1151
Age, Customized [Mean (Full Range); unit: years]
  Age | 87.51 [73 to 102] | 87.22 [66 to 98] | 65 [29 to 96] | 64 [36 to 96] | 47 [20 to 66] | 47 [20 to 65] | 53.77 [37 to 67] | 47 [26 to 66] | 53 [20 to 102]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Age was not given by all participants.
  Participants
    number analyzed (Participants) | 42 | 40 | 152 | 156 | 357 | 330 | 20 | 48 | 1145
    Female | 28 | 24 | 112 | 124 | 333 | 320 | 20 | 44 | 1005
    Male | 14 | 16 | 40 | 32 | 24 | 10 | 0 | 4 | 140
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization Quality of Life-BREF (WHOQOL-BREF)
Description: World Health Organization Quality of Life-BREF (WHOQOL-BREF) measure quality of life for older persons' at the end of life living in nursing homes.
  Five-point Likert-scale. Higher values mean better outcomes. Total score Min 26. Max 130.
  The range for the sub scale Overall Quality of Life; Min 1 Max 5 The range for the sub scale General health; Min 1 Max 5 The range for the sub scale Physical Health; Min 7 Max 35 The range for the sub scale Psychological; Min 6 Max 30 The range for the sub scale Social relationships; Min 3 Max 15 The range for the sub scale Environment; Min 8 Max 40
Time Frame: 9 months
Population: The inclusion criteria for the older persons were that they were 65 years or older, spoke Swedish, did not have dementia and had enough energy to participate in a structured interview for up to one hour.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group Older People | Control Group Older People
Number analyzed (Participants) | 23 | 29
score on a scale
  Total score | 86 [74 to 95] | 82 [77.5 to 90]
  Overall Quality of Life | 3 [2 to 4] | 3 [2.5 to 4]
  General health | 3 [2 to 4] | 3 [2.5 to 4]
  Physical Health | 21 [18 to 25] | 20 [17 to 24.5]
  Psychological | 21 [21 to 23] | 20 [18 to 21.5]
  Social relationships | 8 [7 to 8] | 8 [7.5 to 9]
  Environment | 28 [25 to 33] | 29 [26 to 31]

2. Primary Outcome: World Health Organization Quality of Life-OLD (WHOQOL-OLD)
Description: World Health Organization Quality of Life-OLD (WHOQOL-OLD) measure quality of life for older persons living in nursing homes.
  Five point Likert-scale. Higher value means better outcome. Min 24. Max. 120. The range for the all the sub scales are; Min 1 Max 20
Time Frame: 9 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group Older People | Control Group Older People
Number analyzed (Participants) | 23 | 29
score on a scale
  Sensory Abilities | 15 [12 to 17] | 13 [11 to 15.5]
  Autonomy | 11 [10 to 15] | 12 [10 to 13]
  Past, present and future abilities | 14 [11 to 15] | 14 [12 to 15]
  Social participation | 12 [9 to 16] | 13 [10 to 14]
  Death and Dying | 17 [14 to 19] | 18 [15 to 19]
  Intimacy | 14 [12 to 16] | 14 [12 to 16]

3. Primary Outcome: Person-centred Care Assessment Tool (P-CAT)(Patient Version)
Description: Person-centred Care Assessment Tool (P-CAT) (patient version) measure person-centred care for older persons living in nursing homes. Five point Likert-scale. Higher score means better outcomes. Min 13. Max. 65.
  The range for the sub scale Extent of personalizing care; Min 8 Max 40 The range for the sub scale Amount of organizational and environmental support; Min 5 Max 25
Time Frame: 9 months
Population: In total, 90 older persons, (65 years or older) were included in the study based on the inclusion criteria of being Swedish speaking, not having dementia and with enough energy to manage a structured interview lasting up to one hour.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group Older People | Control Group Older People
Number analyzed (Participants) | 24 | 20
score on a scale
  Extent of personalizing care | 25.0 [18.0 to 32.0] | 27 [22.2 to 29.8]
  Amount of organizational and environmental support | 11.0 [6.5 to 16.5] | 11.0 [10.0 to 16.0]

4. Primary Outcome: Person-Centred Climate Questionnaire (PCQ Patient Version)
Description: Person-Centred Climate Questionnaire (PCQ patient version) measure person-centred care for older persons living in nursing homes. Six point Likert-scale. Higher score means better outcome. Min 17. Max. 102.
  The range for the sub scale Safety; Min 10 Max 60 The range for the sub scale Everydayness; Min 4 Max 24 The range for the sub scale Hospitality; Min 3 Max 18
Time Frame: 9 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group Older People | Control Group Older People
Number analyzed (Participants) | 24 | 20
score on a scale
  Safety | 51.5 [48.5 to 55.8] | 53.0 [47.5 to 58.0]
  Everydayness | 19.5 [17.0 to 23.0] | 19.5 [18.0 to 22.0]
  Hospitality | 15.0 [14.0 to 16.0] | 15.5 [14.2 to 17.0]

5. Primary Outcome: Next-of-Kin Participation in Care (NoK-PiC); Psychometric Evaluation
Description: Next-of-Kin Participation in Care (NoK-PiC) measure participation for next of kin to older persons in nursing homes. The study includes both intervention and control groups. The two scales are 1) Communication and Trust (CaT); and 2) Collaboration in Care (CiC).
  The scales contains nine items each and items are scored from 0 to 4 (agree not at all (=0); agree to a low degree (=1); agree partly (=2); agree to a high degree (=3); and agree totally (=4). The possible score range from 0 to 36 in each of the two scales, and from 0-72 in the total scale. Higher score means better outcomes. This results are based upon a recently published psychometric evaluation by Westergren et al (2020).
Time Frame: 9 months
Population: The inclusion criterion was someone who had a relation to one of the older persons living at the participating nursing homes but not necessarily family members or relatives.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group Next-of-Kin | Control Group Next-of-kin
Number analyzed (Participants) | 95 | 108
score on a scale
  Next-of-Kin Participation in Care | 48.9 (14.9) | 48.6 (14.1)
  Communication and Trust | 27.6 (7.2) | 27.9 (6.6)
  Collaboration in Care | 21.4 (8.6) | 20.7 (8.8)

6. Primary Outcome: World Health Organization Quality of Life-BREF (WHOQOL-BREF) for Next of Kin
Description: World Health Organization Quality of Life-BREF (WHOQOL-BREF) measure quality of life for next of kin to older persons in nursing homes. Five-point Likert-scale. Higher values mean better outcomes. Min 26. Max 130.
  he range for the sub scale Overall Quality of Life; Min 1 Max 5 The range for the sub scale General health; Min 1 Max 5 The range for the sub scale Physical Health; Min 7 Max 35 The range for the sub scale Psychological; Min 6 Max 30 The range for the sub scale Social relationships; Min 3 Max 15 The range for the sub scale Environment; Min 8 Max 40
Time Frame: 9 months
Population: The inclusion criteria were a next of kin who had a relation to an older person living in one of the participating nursing homes but was not necessarily a family member or a relative [14]. The next of kin were recruited consecutively in equal numbers from both the intervention nursing homes and the control nursing homes.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group Next-of-Kin | Control Group Next-of-kin
Number analyzed (Participants) | 90 | 105
score on a scale
  Total score | 94 [87 to 102] | 103 [96 to 111]
  Overall Quality of Life | 4 [4 to 5] | 4 [4 to 5]
  General health | 4 [3 to 4] | 4 [3 to 5]
  Physical Health | 16 [15 to 18] | 16 [14 to 18]
  Psychological | 16 [14 to 17] | 17 [15 to 18]
  Social relationships | 4 [4 to 5] | 4 [4 to 5]
  Environment | 16 [15 to 18] | 17 [15 to 18]

7. Secondary Outcome: Person-centred Care Assessment Tool (P-CAT) (Staff Version)
Description: Person-centred Care Assessment Tool (P-CAT)(staff version) measure person-centred care for staff working in nursing homes. Five-point Likert-scale. Higher values mean better outcomes. Min 13. Max 65.
  The range for the sub scale Extent of personalizing care; Min 8 Max 40 The range for the sub scale Amount of organizational and environmental support; Min 5 Max 25
Time Frame: 6 months
Population: The informants in this study, the staff, were recruited consecutively in equal numbers from both the intervention nursing homes and the control nursing homes.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group Staff | Control Group Staff
Number analyzed (Participants) | 167 | 198
score on a scale
  Total score | 45.0 [42.0 to 48.0] | 44.0 [41.0 to 48.0]
  Extent of personalizing care | 34.0 [32.0 to 37.0] | 34.0 [31.0 to 36.0]
  Amount of organizational and environmental support | 11.0 [8.0 to 14.0] | 11.0 [8.0 to 15.0]

8. Secondary Outcome: Person-Centred Climate Questionnaire (PCQ-S)
Description: Person-Centred Climate Questionnaire (PCQ-S) measure person-centred care for staff working in nursing homes. Six-point Likert-scale. Higher values mean better outcomes. Min 14. Max 84.
  The range for the sub scale Safety; Min 5 Max 30 The range for the sub scale Everydayness; Min 5 Max 30 The range for the sub scale Community; Min 4 Max 24
Time Frame: 6 months
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention Group Staff | Control Group Staff
Number analyzed (Participants) | 167 | 198
score on a scale
  Total score | 77.0 [68.0 to 81.0] | 74.0 [67.0 to 79.0]
  Safety | 27.0 [25.0 to 30.0] | 27.0 [24.0 to 29.0]
  Everydayness | 25.0 [22.0 to 29.0] | 25.0 [21.0 to 27.0]
  Community | 23.0 [20.0 to 24.0] | 22.0 [21.0 to 24.0]

ADVERSE EVENTS:
Time Frame: Data were collected at baseline and three months after the intervention was completed i.e nine months after baseline. Phase one data collection began 25th April 2015 and ended 31st March 2016. Phase two data collection began 23th August 2016 and ended 17th June 2017. After the main data collection period, there were a few (3) interviews missing with managers which were conducted until 15 October 2017.
Description: Due to major drop-outs among older people (death) and staff (limited time) the cross-over design was not possible to fulfilled as planned from the start of the project (see more details in the study protocol).
Groups:
- Intervention Group Older People; Control Group Older People: Older persons: The inclusion criteria for the older persons were ≥ 65 years without dementia, speaking Swedish and with enough energy to manage a structured interview during up to one hour.
- Intervention Group Next of Kin; Control Group Next of Kin: The inclusion criterion was someone who had a relation to one of the older persons living at the participating nursing homes but not necessarily family members or relatives.
- Intervention Group Staff; Control Group Staff: The inclusion criterion was staff at nursing homes (commonly assistant nurses, nurses, occupational therapists and physiotherapists).
- Intervention Group Managers: Managers at different levels with responsibility for the care and social service at the included nursing homes
Arm/Group | Intervention Group Older People | Control Group Older People | Intervention Group Next of Kin | Control Group Next of Kin | Intervention Group Staff | Control Group Staff | Intervention Group Managers | Intervention Focus Groups Staff
All-Cause Mortality (participants affected / at risk) | 20/42 | 19/40 | 0/152 | 0/156 | 1/363 | 0/330 | 0/20 | 0/48
Serious Adverse Events (participants affected / at risk) | 20/42 | 19/40 | 0/152 | 0/156 | 1/363 | 0/330 | 0/20 | 0/48
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40 | 62/152 | 51/156 | 195/363 | 132/330 | 0/20 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group Older People (N=42) | Control Group Older People (N=40) | Intervention Group Next of Kin (N=152) | Control Group Next of Kin (N=156) | Intervention Group Staff (N=363) | Control Group Staff (N=330) | Intervention Group Managers (N=20) | Intervention Focus Groups Staff (N=48)
Death (General disorders) | 20 (20) | 19 (19) | NA | NA | 1 (1) | NA | NA | NA — Frailty and old age (not related to the intervention)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group Older People (N=42) | Control Group Older People (N=40) | Intervention Group Next of Kin (N=152) | Control Group Next of Kin (N=156) | Intervention Group Staff (N=363) | Control Group Staff (N=330) | Intervention Group Managers (N=20) | Intervention Focus Groups Staff (N=48)
Other (Social circumstances) | 0 (0) | 0 (0) | 62 (152) | 51 (156) | 195 (363) | 132 (330) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT02708498/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT02708498/SAP_003.pdf